CLINICAL TRIAL: NCT04896866
Title: Efficacy and Safety of Antimicrobial Stewardship Intervention in Hospitalized COVID-19 Patients: A Pragmatic Clinical Trial
Brief Title: Efficacy and Safety of Antimicrobial Stewardship Intervention in Hospitalized COVID-19 Patients (COVASP)
Acronym: COVASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00105598
Record Dates: First submitted 2021-05-17; First posted 2021-05-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-04

CONDITIONS: Covid19; COVID-19 Pneumonia; COVID-19 Lower Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome; SARS-CoV2 Infection; SARS-CoV-2 Acute Respiratory Disease
Keywords: antimicrobial stewardship; antibiotic stewardship; prospective audit and feedback; quality improvement; antibiotics
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Hospital beds are randomized prior to enrolment to intervention versus observation. Intervention consists of antimicrobial stewardship prospective audit and feedback.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antimicrobial stewardship (Experimental): Antimicrobial stewardship prospective audit and feedback on physicians attending to patients admitted with community-acquired COVID-19 pneumonia to beds randomized to antimicrobial stewardship intervention.
  Interventions: Behavioral: Antimicrobial stewardship prospective audit and feedback
- No antimicrobial stewardship (No Intervention): No antimicrobial stewardship prospective audit and feedback.

INTERVENTIONS:
Behavioral: Antimicrobial stewardship prospective audit and feedback — Audits are performed on weekdays, less statutory holidays, by members of the antimicrobial stewardship team consisting of infectious disease or antimicrobial stewardship physicians or pharmacists. Verbal and written feedback will be provided in real-time. Initial prospective audit and feedback (PAF) will occur on the day of enrolment. Follow-up PAF will occur weekly (+/-3 days to account for weekends or statuary holidays) and ad-hoc if a new antibacterial is prescribed, until the primary end-point. Appropriateness will be assessed based on local clinical practice guidelines. Only antibacterials will be audited. Prescriptions will be excluded from PAF if they are single doses or discontinued prior to PAF. Prescriptions will be also be excluded from PAF and the final analysis if being used for surgical or medical prophylaxis.
  Arms: Antimicrobial stewardship

SUMMARY:
COVID-19 is respiratory disease caused by the severe acute respiratory coronavirus 2 (SARS-CoV-2), a novel coronavirus which has spread rapidly across the world with over 149.9 million laboratory confirmed cases and over 3.1 million reported deaths since December 2019. Approximately 4-8% of hospitalized patients with COVID-19 have co-infection with bacterial pathogens however there is widespread and often broad-spectrum antibiotic use in these patients.

This is a prospective, multi-center, non-inferiority pragmatic clinical trial of antimicrobial stewardship prospective audit and feedback versus no antimicrobial stewardship intervention on physicians attending to patients with proven SARS-CoV-2 infection confirmed by nucleic acid testing in the preceding 2 weeks of hospitalization for acute COVID-19 pneumonia. Prospective audit and feedback is the real time review of antibacterial prescriptions and immediate feedback to prescribers to optimize antimicrobial prescriptions. Hospital beds will be stratified by COVID unit and critical care unit beds, and will be computer randomized in a 1:1 fashion into 2 arms (antimicrobial stewardship intervention versus no antimicrobial stewardship intervention) prior to study commencement at the participating site. Patients hospitalized to study-eligible beds will be followed for primary and secondary outcomes.

The objective of this study is to determine the effect of an antimicrobial stewardship intervention (prospective audit and feedback) on clinical outcomes in patients hospitalized with acute COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of hospital admission.
* Confirmed SARS-CoV-2 infection by nucleic acid testing in the preceding 14 days of hospital admission.
* Admitted from the community (including continuing care facilities).
* Admitted to a hospital bed designated in the study.
* SpO2 ≤94% requiring supplemental oxygen or chest imaging findings compatible with COVID-19 pneumonia.

Exclusion Criteria:

* The patient is enrolled in another clinical trial that involves antibacterial therapy.
* The patient's goals of care is anticipated to be designated "total compassionate care" or palliative care within 48 hours of admission.
* The patient's progression to death is anticipated to be imminent and inevitable within 48 hours of admission.
* The patient was attended by any member of the research team within 30 days of enrollment.
* The patient is transferred from another acute care center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Ordinal scale | Day 15 of hospital admission
  A 7 point ordinal scale of clinical outcomes:
  1. point - Not hospitalized, able to resume normal daily activities
  2. points - Not hospitalized, unable to resume normal daily activities
  3. points - Hospitalized, not on supplemental oxygen
  4. points - Hospitalized, on supplemental oxygen
  5. points - Hospitalized, on high flow oxygen therapy or non-invasive mechanical ventilation
  6. points - Hospitalized, on ECMO or invasive mechanical ventilation
  7. points - Death
  Higher scores means a worse outcome.

SECONDARY OUTCOMES:
Length of hospital stay | through study completion, an average of 5 days
  Duration of hospitalization in days
In-hospital mortality | through study completion, an average of 5 days
  Death occurring during hospital admission
30-day mortality | 30 days
  Mortality in the first 30 days after diagnosis
30-day C. difficile associated mortality | 30 days
  Death related to C. difficile-associated diarrhea in the first 30 days after diagnosis
30 day re-admission rate | 30 days from hospital discharge
  Re-admission to hospital after initial discharge in the first 30 days after diagnosis
Days of therapy normalized for patient-days | capped at 30 days of hospitalization
  Days of antibiotic therapy normalized for patients-day
Length of total antimicrobial therapy normalized for patient-days | capped at 30 days of hospitalization
  Length of antibiotics normalized for patient-days
Number of antimicrobial stewardship audits | through study completion, an average of 5 days
  Number of audits by ASP
Number of antimicrobial stewardship recommendations | through study completion, an average of 5 days
  Number of recommendations by ASP
Antimicrobial stewardship acceptance rates | through study completion, an average of 5 days
  Acceptance rate of ASP recommendations
Multi-drug resistant bacteria infection rates | 30 days
  Development of multi-drug resistant bacterial infection in the first 30 days after diagnosis
Clostridioides difficile infection rate | 30 days
  C. difficile-associated diarrhea in the first 30 days after diagnosis
Percentage of participants with neutropenia | 30 days
  Occurrence of neutropenia in the first 30 days
Acute kidney injury | 30 days
  diagnosed and staged as according to KDIGO

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Misericordia Community Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published in an open journal.
Supporting Information: Study Protocol

REFERENCES:
- [Background] MacIntyre CR, Chughtai AA, Barnes M, Ridda I, Seale H, Toms R, Heywood A. The role of pneumonia and secondary bacterial infection in fatal and serious outcomes of pandemic influenza a(H1N1)pdm09. BMC Infect Dis. 2018 Dec 7;18(1):637. doi: 10.1186/s12879-018-3548-0. PMID 30526505
- [Background] Shah NS, Greenberg JA, McNulty MC, Gregg KS, Riddell J 4th, Mangino JE, Weber DM, Hebert CL, Marzec NS, Barron MA, Chaparro-Rojas F, Restrepo A, Hemmige V, Prasidthrathsint K, Cobb S, Herwaldt L, Raabe V, Cannavino CR, Hines AG, Bares SH, Antiporta PB, Scardina T, Patel U, Reid G, Mohazabnia P, Kachhdiya S, Le BM, Park CJ, Ostrowsky B, Robicsek A, Smith BA, Schied J, Bhatti MM, Mayer S, Sikka M, Murphy-Aguilu I, Patwari P, Abeles SR, Torriani FJ, Abbas Z, Toya S, Doktor K, Chakrabarti A, Doblecki-Lewis S, Looney DJ, David MZ. Bacterial and viral co-infections complicating severe influenza: Incidence and impact among 507 U.S. patients, 2013-14. J Clin Virol. 2016 Jul;80:12-9. doi: 10.1016/j.jcv.2016.04.008. Epub 2016 Apr 14. PMID 27130980
- [Background] Rawson TM, Moore LSP, Zhu N, Ranganathan N, Skolimowska K, Gilchrist M, Satta G, Cooke G, Holmes A. Bacterial and Fungal Coinfection in Individuals With Coronavirus: A Rapid Review To Support COVID-19 Antimicrobial Prescribing. Clin Infect Dis. 2020 Dec 3;71(9):2459-2468. doi: 10.1093/cid/ciaa530. PMID 32358954
- [Background] Langford BJ, So M, Raybardhan S, Leung V, Westwood D, MacFadden DR, Soucy JR, Daneman N. Bacterial co-infection and secondary infection in patients with COVID-19: a living rapid review and meta-analysis. Clin Microbiol Infect. 2020 Dec;26(12):1622-1629. doi: 10.1016/j.cmi.2020.07.016. Epub 2020 Jul 22. PMID 32711058
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Feng Y, Ling Y, Bai T, Xie Y, Huang J, Li J, Xiong W, Yang D, Chen R, Lu F, Lu Y, Liu X, Chen Y, Li X, Li Y, Summah HD, Lin H, Yan J, Zhou M, Lu H, Qu J. COVID-19 with Different Severities: A Multicenter Study of Clinical Features. Am J Respir Crit Care Med. 2020 Jun 1;201(11):1380-1388. doi: 10.1164/rccm.202002-0445OC. PMID 32275452
- [Background] Wan S, Xiang Y, Fang W, Zheng Y, Li B, Hu Y, Lang C, Huang D, Sun Q, Xiong Y, Huang X, Lv J, Luo Y, Shen L, Yang H, Huang G, Yang R. Clinical features and treatment of COVID-19 patients in northeast Chongqing. J Med Virol. 2020 Jul;92(7):797-806. doi: 10.1002/jmv.25783. Epub 2020 Apr 1. PMID 32198776
- [Background] Wang Z, Yang B, Li Q, Wen L, Zhang R. Clinical Features of 69 Cases With Coronavirus Disease 2019 in Wuhan, China. Clin Infect Dis. 2020 Jul 28;71(15):769-777. doi: 10.1093/cid/ciaa272. PMID 32176772
- [Background] Zhao XY, Xu XX, Yin HS, Hu QM, Xiong T, Tang YY, Yang AY, Yu BP, Huang ZP. Clinical characteristics of patients with 2019 coronavirus disease in a non-Wuhan area of Hubei Province, China: a retrospective study. BMC Infect Dis. 2020 Apr 29;20(1):311. doi: 10.1186/s12879-020-05010-w. PMID 32345226
- [Background] Cao J, Hu X, Cheng W, Yu L, Tu WJ, Liu Q. Clinical features and short-term outcomes of 18 patients with corona virus disease 2019 in intensive care unit. Intensive Care Med. 2020 May;46(5):851-853. doi: 10.1007/s00134-020-05987-7. Epub 2020 Mar 2. No abstract available. PMID 32123993
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Barrasa H, Rello J, Tejada S, Martin A, Balziskueta G, Vinuesa C, Fernandez-Miret B, Villagra A, Vallejo A, San Sebastian A, Cabanes S, Iribarren S, Fonseca F, Maynar J; Alava COVID-19 Study Investigators. SARS-CoV-2 in Spanish Intensive Care Units: Early experience with 15-day survival in Vitoria. Anaesth Crit Care Pain Med. 2020 Oct;39(5):553-561. doi: 10.1016/j.accpm.2020.04.001. Epub 2020 Apr 9. PMID 32278670
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Du Y, Tu L, Zhu P, Mu M, Wang R, Yang P, Wang X, Hu C, Ping R, Hu P, Li T, Cao F, Chang C, Hu Q, Jin Y, Xu G. Clinical Features of 85 Fatal Cases of COVID-19 from Wuhan. A Retrospective Observational Study. Am J Respir Crit Care Med. 2020 Jun 1;201(11):1372-1379. doi: 10.1164/rccm.202003-0543OC. PMID 32242738
- [Background] Polgreen PM, Chen YY, Cavanaugh JE, Ward M, Coffman S, Hornick DB, Diekema DJ, Herwaldt LA. An outbreak of severe Clostridium difficile-associated disease possibly related to inappropriate antimicrobial therapy for community-acquired pneumonia. Infect Control Hosp Epidemiol. 2007 Feb;28(2):212-4. doi: 10.1086/512174. Epub 2007 Jan 25. PMID 17265406
- [Background] Sapp JL, Alqarawi W, MacIntyre CJ, Tadros R, Steinberg C, Roberts JD, Laksman Z, Healey JS, Krahn AD. Guidance on Minimizing Risk of Drug-Induced Ventricular Arrhythmia During Treatment of COVID-19: A Statement from the Canadian Heart Rhythm Society. Can J Cardiol. 2020 Jun;36(6):948-951. doi: 10.1016/j.cjca.2020.04.003. Epub 2020 Apr 8. PMID 32299753
- [Background] Clancy CJ, Nguyen MH. Coronavirus Disease 2019, Superinfections, and Antimicrobial Development: What Can We Expect? Clin Infect Dis. 2020 Dec 17;71(10):2736-2743. doi: 10.1093/cid/ciaa524. PMID 32361747
- [Background] Stevens MP, Patel PK, Nori P. Involving antimicrobial stewardship programs in COVID-19 response efforts: All hands on deck. Infect Control Hosp Epidemiol. 2020 Jun;41(6):744-745. doi: 10.1017/ice.2020.69. No abstract available. PMID 32167442
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Derived] Chen JZ, Hoang HL, Yaskina M, Kabbani D, Doucette KE, Smith SW, Lau C, Stewart J, Remtulla S, Zurek K, Schultz M, Koriyama-McKenzie H, Cervera C. Efficacy and safety of antimicrobial stewardship prospective audit and feedback in patients hospitalised with COVID-19 (COVASP): a pragmatic, cluster-randomised, non-inferiority trial. Lancet Infect Dis. 2023 Jun;23(6):673-682. doi: 10.1016/S1473-3099(22)00832-5. Epub 2023 Jan 27. PMID 36716763
- [Derived] Chen JZ, Hoang HL, Yaskina M, Kabbani D, Doucette KE, Smith SW, Lau C, Stewart J, Zurek K, Schultz M, Cervera C. Efficacy and safety of antimicrobial stewardship prospective audit and feedback in patients hospitalized with COVID-19: A protocol for a pragmatic clinical trial. PLoS One. 2022 Mar 23;17(3):e0265493. doi: 10.1371/journal.pone.0265493. eCollection 2022. PMID 35320289